CLINICAL TRIAL: NCT02154399
Title: Pilot Phase II Research Study of EF5 to Measure Tumor Hypoxia in Patients With Non-small Cell Lung Cancer
Brief Title: EF5 in Measuring Tumor Hypoxia in Patients With Stage I-III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01169; NCI-2014-01169 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2310 (Other: Duke University Medical Center); 2310 (Other: CTEP); P30CA014236 (NIH); R21CA091565 (NIH)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2014-06

CONDITIONS: Stage IA Non-Small Cell Lung Carcinoma; Stage IB Non-Small Cell Lung Carcinoma; Stage IIA Non-Small Cell Lung Carcinoma; Stage IIB Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (EF5) (Experimental): Patients receive EF5 IV over 1-2.5 hours. Beginning 24-55 hours later, patients undergo tumor hypoxia measurement using a polarographic needle electrode and intraoperative tumor measurement before undergoing surgical biopsy or resection.
  Interventions: Drug: EF5; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery; Other: Tissue Oxygen Measurement

INTERVENTIONS:
Drug: EF5 — Given IV
  Other Names: EF-5
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery/thoracotomy
Other: Tissue Oxygen Measurement — Undergo tumor hypoxia measurement

SUMMARY:
This pilot phase II trial studies how well EF5 works in measuring lack of tumor oxygen, hypoxia, in patients with stage I-III non-small cell lung cancer. EF5 may be effective in measuring the lack of oxygen in lung tumors and may allow doctors to plan better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the frequency and degree of hypoxia as measured by EF5 binding in patients with non-small cell lung cancer.

II. Correlate hypoxia as measured by EF5 binding with potential serum/plasma markers of hypoxia in patients with non-small cell lung cancer.

III. Correlate hypoxia as measured by EF5 binding with tissue markers of hypoxia in patients with non-small cell lung cancer.

IV. Correlate hypoxia as measured by EF5 binding with tumor angiogenesis in patients with non-small cell lung cancer.

V. Correlated hypoxia as measured by EF5 binding with apoptosis in patients with non-small cell lung cancer.

VI. Measure and characterize tumor perfusion in relationship to hypoxia in patients with non-small cell lung cancer.

VII. Correlate tumor perfusion to microvessel density in tumor samples in patients with non-small cell lung cancer.

VIII. Determine the longevity of EF5 adducts in human lung tumors.

OUTLINE:

Patients receive EF5 intravenously (IV) over 1-2.5 hours. Beginning 24-55 hours later, patients undergo tumor hypoxia measurement using a polarographic needle electrode and intraoperative tumor measurement before undergoing surgical biopsy or resection.

After completion of study treatment, patients are followed up for 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected non-small cell lung cancer; patients without histologically or cytologically documented non-small cell lung cancer (NSCLC) must be estimated by their physician to have at least 75% probability of having NSCLC; the probability of malignancy will be predicted on the basis of known probabilities of individual clinical characteristics using a Bayesian model
* Clinical or pathologic stage I to III; patients in whom pre-surgical staging has not definitively establish stage IV disease are eligible
* Tumor mass at least 1.5 cm in maximum diameter must be present on computed tomography (CT) scan and must be included in the planned surgical biopsy or resection
* Patient must be planning to undergo a surgical staging or treatment procedure (including mediastinoscopy, wedge resection, lobectomy, or pneumonectomy) and have the clinical and physiological status appropriate for this procedure
* Performance status 0-2
* Bilirubin within normal limits
* Creatinine within normal limits or, if elevated, a creatinine clearance of at least 60 mL/min/m^2 (EF5 is primarily excreted via the kidney)
* White blood cell (WBC) > 2000/mm^3
* Platelets > 100,000/mm^3

Exclusion Criteria:

* Pregnancy or breast feeding; a negative serum pregnancy test is required of any woman of childbearing potential prior to enrollment; pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with EF5
* Allergy to IV contrast dye
* History of grade III or IV peripheral neuropathy as defined by the National Cancer Institute (NCI) Common Terminology Criteria (CTC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-05; Primary Completion 2007-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Frequency and degree of hypoxia using a polarographic needle electrode | 55 hours post-EF5 infusion
Serum/plasma markers of hypoxia | 55 hours post-EF5 infusion
  Spearman's rank correlation will be used to examine the relationship between hypoxia as measured by EF5 binding with serum markers of hypoxia (vascular endothelial growth factor [VEGF], D-Dimer, plasminogen activator inhibitor type 1 [PAI-1]).
Tissue markers of hypoxia | 55 hours post-EF5 infusion
  Spearman's rank correlation will be used to examine the relationship between hypoxia as measured by EF5 binding with tissue markers of hypoxia (hypoxia inducible factor 1 [HIF-1] alpha, involucrin).
Tumor perfusion using dynamic positron emission tomography | 10 days prior to surgery
  Spearman's rank correlation will be used to examine the relationship between hypoxia as measured by EF5 binding with tumor perfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kelley, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Durham Veterans Affairs Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina